CLINICAL TRIAL: NCT05763316
Title: Accuracy of Scoring Systems for Risk Assessment in Neonatal Intensive Care Unit at Sohag University Hospital
Brief Title: Accuracy of Scoring Systems for Risk Assessment in Neonatal Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rehab Zain Elabdeen Abdelfattah, Pediatric Resident, Sohag University
Other Study IDs: Soh-Med-23-03-10MS
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Neonatal Death
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study participants: Neonates admitted to NICU and fulfilling eligibility criteria
  Interventions: Other: CRIB II; Other: SNAP-II; Other: SNAPPE-II; Other: STOPS; Other: MSNS; Other: nSOFA

INTERVENTIONS:
Other: CRIB II — Calculate Clinical Risk Index for Babies II score
Other: SNAP-II — Calculate Score for Neonatal Acute Physiology II
Other: SNAPPE-II — Calculate Score for Neonatal Acute Physiology Perinatal Extension II
Other: STOPS — Calculate Sensorium, temperature, oxygenation, perfusion, skin color, and blood sugar score
Other: MSNS — Calculate Modified Sick neonatal Score
Other: nSOFA — Calculate neonatal sequential organ failure assessment

SUMMARY:
Early detection of neonates with higher risk of death is quite important for paying more attention to these cases, timely referral to tertiary neonatal intensive care unit (NICU), and provision of meticulous critical care, which ultimately may improve outcomes. Several scoring systems have recently been developed for assessment of the intensity of illness and prognosticate the risk of not only neonatal mortality but also short- and long-term morbidities. The accuracy of these scoring systems has been investigated in several NICUs from different countries, such as USA, UK, Canada, Brazil, India, and Iran. Previous Egyptian studies have investigated the accuracy of Clinical Risk Index for Babies II (CRIB II), Score for Neonatal Acute Physiology II (SNAP-II) and its Perinatal Extension II (SNAPPE-II). However, the accuracy of Sensorium, temperature, oxygenation, perfusion, skin color, and blood sugar (STOPS), Modified Sick neonatal Score (MSNS), and neonatal sequential organ failure assessment (nSOFA) has not been investigated in Egyptian NICUs. Therefore, more studies are required to investigate the utility and accuracy of neonatal risk assessment scores in Egyptian NICUs.

ELIGIBILITY:
Inclusion Criteria:

* Admission within 24 hours after birth.
* Length of hospital stay at the first admission to NICU ≥12 hours

Exclusion Criteria:

* Major congenital anomalies.
* Discharge against medical advice
* Transportation to other places.
* Missing data on items of scoring systems

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates admitted to NICUs at Sohag University Hospitals during the study duration
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-12 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Survival at discharge | One year
  Proportion of neonates discharged alive from NICU

SECONDARY OUTCOMES:
Length of hospital stay | One year
  Length of stay in NICU
Need for CPAP | One year
  Proportion of neonates connected to continuous positive airway pressure
Need for invasive ventilation | One year
  Proportion of neonates requiring invasive ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Montaser M Mohamed, MD, PhD, Study Chair — Sohag University
Locations (1):
- Neonatal Intensive Care Units at Sohag University Hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual participant data will be available from the principal investigator upon a reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: After publication and for three years
Access Criteria: Available from the principal investigator upon a reasonable request

REFERENCES:
- [Background] Garg B, Sharma D, Farahbakhsh N. Assessment of sickness severity of illness in neonates: review of various neonatal illness scoring systems. J Matern Fetal Neonatal Med. 2018 May;31(10):1373-1380. doi: 10.1080/14767058.2017.1315665. Epub 2017 Apr 20. PMID 28372507
- [Background] Vardhelli V, Murki S, Tandur B, Saha B, Oleti TP, Deshabhotla S, Mohammed YA, Seth S, Siramshetty S, Kallem VR. Comparison of CRIB-II with SNAPPE-II for predicting survival and morbidities before hospital discharge in neonates with gestation </= 32 weeks: a prospective multicentric observational study. Eur J Pediatr. 2022 Jul;181(7):2831-2838. doi: 10.1007/s00431-022-04463-2. Epub 2022 May 6. PMID 35524143
- [Background] Parry G, Tucker J, Tarnow-Mordi W; UK Neonatal Staffing Study Collaborative Group. CRIB II: an update of the clinical risk index for babies score. Lancet. 2003 May 24;361(9371):1789-91. doi: 10.1016/S0140-6736(03)13397-1. PMID 12781540
- [Background] Richardson DK, Corcoran JD, Escobar GJ, Lee SK. SNAP-II and SNAPPE-II: Simplified newborn illness severity and mortality risk scores. J Pediatr. 2001 Jan;138(1):92-100. doi: 10.1067/mpd.2001.109608. PMID 11148519
- [Background] Vardhelli V, Seth S, Mohammed YA, Murki S, Tandur B, Saha B, Oleti TP, Deshabhotla S, Siramshetty S, Kallem VR. Comparison of STOPS and SNAPPE-II in Predicting Neonatal Survival at Hospital Discharge: A Prospective, Multicentric, Observational Study. Indian J Pediatr. 2023 Aug;90(8):781-786. doi: 10.1007/s12098-022-04330-w. Epub 2022 Sep 22. PMID 36136230
- [Background] Mansoor KP, Ravikiran SR, Kulkarni V, Baliga K, Rao S, Bhat KG, Baliga BS, Kamath N. Modified Sick Neonatal Score (MSNS): A Novel Neonatal Disease Severity Scoring System for Resource-Limited Settings. Crit Care Res Pract. 2019 May 9;2019:9059073. doi: 10.1155/2019/9059073. eCollection 2019. PMID 31210987
- [Background] Wynn JL, Polin RA. A neonatal sequential organ failure assessment score predicts mortality to late-onset sepsis in preterm very low birth weight infants. Pediatr Res. 2020 Jul;88(1):85-90. doi: 10.1038/s41390-019-0517-2. Epub 2019 Aug 8. PMID 31394566
- [Background] Ezz-Eldin ZM, Hamid TA, Youssef MR, Nabil Hel-D. Clinical Risk Index for Babies (CRIB II) Scoring System in Prediction of Mortality in Premature Babies. J Clin Diagn Res. 2015 Jun;9(6):SC08-11. doi: 10.7860/JCDR/2015/12248.6012. Epub 2015 Jun 1. PMID 26266178